CLINICAL TRIAL: NCT02694900
Title: Comparison of Three Different Chest Compressions Methods During Pediatric Cardiopulmonary Resuscitation: A Pilot, Randomized Crossover Manikin Trial
Brief Title: Single-rescuer Pediatric Resuscitation
Acronym: SRPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02.009.1MR
Record Dates: First submitted 2016-02-16; First posted 2016-03-01 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Chest Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resuscitation on the flor (Experimental): 2 min asynchronous cardiopulmonary resuscitation. The patient lies on the floor
  Interventions: Other: Manually chest compressions; Device: Cardiopump; Device: LifeLine ARM
- Resuscitation on the stretcher (Experimental): 2 min asynchronous cardiopulmonary resuscitation. The patient lies on a stretcher
  Interventions: Other: Manually chest compressions; Device: Cardiopump; Device: LifeLine ARM

INTERVENTIONS:
Other: Manually chest compressions — Chest compressions performed manually without any device
Device: Cardiopump — Chest compressions performed with Cardiopump
Device: LifeLine ARM — Chest compressions performed using mechanical chest compressions system LifeLine ARM

SUMMARY:
The objective of this pilot study was to compare the manual chest compressions (CC) versus CC feedback device TrueCPR vs mechanical CC device LifeLine ARM during simulated pediatric cardiopulmonary resuscitation

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* maximum 1 year of work experience in medicine
* minimum 10 clinical resuscitations
* paramedics, nurses, physicians

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
chest compressions effectiveness | 1 day
  the percentage of correct chest compressions relative to the total number of chest compressions

SECONDARY OUTCOMES:
Depth | 1 day
  correct depth according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
Pressure point | 1 day
  correct pressure point according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
Complete pressure release | 1 day
  Complete pressure release measure by manikin software
Rate of chest compressions | 1 day
  correct chest compressions rate according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
Ease-of-use | 1 day
  To access subjective opinion about the difficulty of each chest compression method, participants were asked to rate it on a visual analog scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult).

CONTACTS AND LOCATIONS:
Locations (1):
- Łukasz Szarpak, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Truszewski Z, Szarpak L, Kurowski A, Evrin T, Zasko P, Bogdanski L, Czyzewski L. Randomized trial of the chest compressions effectiveness comparing 3 feedback CPR devices and standard basic life support by nurses. Am J Emerg Med. 2016 Mar;34(3):381-5. doi: 10.1016/j.ajem.2015.11.003. Epub 2015 Nov 4. PMID 26612703